CLINICAL TRIAL: NCT02612493
Title: Obesity and Metabolic Surgery in Patients With Type I Diabetes
Status: Completed | Type: Observational
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Christine Stier, MD, PhD, Sana Klinikum Offenbach
Other Study IDs: FF 120/2015
Record Dates: First submitted 2015-11-17; First posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Type I Diabetes
Keywords: obesity surgery; type I diabetes; weight loss; insulin dosage; postsurgery metabolic changes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Obese patients with type I diabetes — Postsurgical follow - up in obese patients with type I diabetes

SUMMARY:
Obesity is the indication for bariatric surgery in type I diabetes. Interestingly postsurgery the patients improve remarkable in their need for insulin, not only in the daily total insulin dosage but also in the dosage of IU per kg.

DETAILED DESCRIPTION:
The investigators performed a retrospective analysis on 16 patients undergoing weight loss surgery in obesity with concomitant type I diabetes. All patients were evaluated during Follow - Up to analyze insulin dosage and metabolic changes.

ELIGIBILITY:
Inclusion Criteria:

* type I diabetes
* BMI > 40kg/m2

Exclusion Criteria:

* type II diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All obeses patients with type I diabetes who underwent weight loss surgery in our department.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Insulin dosage | up to 8 years
  Insulin dosage postsurgery

SECONDARY OUTCOMES:
Excess Weight loss in % | up to 8 years
Change in HgA1c | up to 8 years
Change in lipids | up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Weiner, MD, Prof., Study Chair — Sana Klinikum Offenbach

REFERENCES:
- [Result] Raab H, Weiner RA, Frenken M, Rett K, Weiner S. Obesity and metabolic surgery in type 1 diabetes mellitus. Nutr Hosp. 2013 Mar;28 Suppl 2:31-4. doi: 10.3305/nh.2013.28.sup2.6711. PMID 23834044
- [Result] Kirwan JP, Brethauer SA, Aminian A, Rosenthal RJ, Kashyap SR, Schauer PR. Response to comments on Brethauer et al. Bariatric surgery improves the metabolic profile of morbidly obese patients with type 1 diabetes. Diabetes care 2014;37:e51-e52. Diabetes Care. 2014 Nov;37(11):e251. doi: 10.2337/dc14-1769. No abstract available. PMID 25342846
- [Result] Brethauer SA, Aminian A, Rosenthal RJ, Kirwan JP, Kashyap SR, Schauer PR. Bariatric surgery improves the metabolic profile of morbidly obese patients with type 1 diabetes. Diabetes Care. 2014;37(3):e51-2. doi: 10.2337/dc13-1736. No abstract available. PMID 24558084